CLINICAL TRIAL: NCT00856258
Title: A Phase 1, Double Blind (Sponsor Open), Randomized, Placebo Controlled, Parallel Group, Oral Multiple Dose Trial To Evaluate The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of PF 03882845 In Healthy Volunteers
Brief Title: Multiple Dose Study in Healthy Volunteers to Assess Safety, Pharmacokinetics and Pharmacodynamics of PF 03882845
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: B0171002
Record Dates: First submitted 2009-03-03; First posted 2009-03-05 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Healthy Volunteers
Keywords: Multiple dose in healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Placebo Comparator): Cohort 1 completed.
  Interventions: Drug: PF 03882845 and Placebo
- Cohort 2 (Placebo Comparator): Cohort 2 not studied
  Interventions: Drug: PF 03882845 and Placebo
- Cohort 3 (Placebo Comparator): Cohort 3 not studied
  Interventions: Drug: PF 03882845 and Placebo
- Cohort 4 (Placebo Comparator): Cohort 4 not studied
  Interventions: Drug: PF 03882845 and Placebo

INTERVENTIONS:
Drug: PF 03882845 and Placebo — The constituted dosage form for all doses were suspensions of drug candidate. Doses were administered once daily for 10 consecutive days.
  Arms: Cohort 1
Drug: PF 03882845 and Placebo — The constituted dosage form for all doses will be suspensions of drug candidate. Doses will be once daily for 10 consecutive days.
  Arms: Cohort 2
Drug: PF 03882845 and Placebo — The constituted dosage form for all doses will be suspensions of drug candidate. Doses will be once daily for 10 consecutive days.
  Arms: Cohort 3
Drug: PF 03882845 and Placebo — The constituted dosage form for all doses will be suspensions of drug candidate. Doses will be once daily for 10 consecutive days.
  Arms: Cohort 4

SUMMARY:
To demonstrate the safety, pharmacokinetics and pharmacodynamics of drug candidate.

DETAILED DESCRIPTION:
The study was terminated on June 19, 2009. Decision to terminate was based on Cohort 1 related safety concerns. An alternative clinical design was envisaged to better assess the benefit to risk.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects of non-childbearing potential between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests.
* An informed consent document signed and dated by the subject or a legally acceptable representative.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant disease, allergy or clinical findings at screening.
* A positive urine drug screen, history of significant regular alcohol consumption within 6 months of screening or use of tobacco or nicotine containing products within the three months preceding study date or a positive urine cotinine at screening or Day -3.
* Blood donation of approximately 1 pint (500 mL) within 56 days prior to dosing.
* Pregnant or nursing females; females of childbearing potential.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Single Dose PK: Cmax, Tmax, and AUCtau; Multiple Dose PK (Assumed Steady State): Cmax(ss), Tmax(ss), AUC(tau,ss), half life, Cmin(ss), Cave(ss), Ae%, CL/F, V/F, CL renal; accumulation ratios AUC(tau,ss)/AUC(tau,sd) and Cmax(ss)/Cmax(sd). | 13 days
Safety and tolerability as determined by adverse event reporting, clinical laboratory results, vital signs (supine blood pressure and heart rate), physical examinations, and electrocardiograms (ECGs). | 13 days

SECONDARY OUTCOMES:
Area under the effect curve (AUEC) for serum aldosterone and plasma renin activity (PRA) on Days 0, 1 and 10. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0171002&StudyName=Multiple%20dose%20study%20in%20healthy%20volunteers%20to%20assess%20safety%2C%20pharmacokinetics%20and%20pharmacodynamics%20of%20PF%2003882845